CLINICAL TRIAL: NCT00034346
Title: A Two Part, Multiple Dose Clinical Trial of the Safety and Efficacy of ABX-EGF in Combination With Paclitaxel and Carboplatin in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: ABX-EGF in Combination With Paclitaxel and Carboplatin for the Treatment of Advanced Non-Small-Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20025404; NCT00068562 (obsolete NCT alias)
Record Dates: First submitted 2002-04-25; First posted 2002-04-26 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Non-Small Cell Lung Cancer; Neoplasm Metastasis; Lung Cancer
Keywords: Advanced; Non-Small-Cell; Lung; Cancer; NSCLC; Carcinoma; Advanced Non-Small-Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms; Neoplasms; Carcinoma | interventions — Panitumumab; Paclitaxel; Carboplatin

INTERVENTIONS:
Drug: ABX-EGF
Drug: paclitaxel
Drug: carboplatin

SUMMARY:
Rationale: Overexpression of epidermal growth factor receptor (EGFR) has been observed in kidney, prostate, colon, lung, breast, and other cancers, and is often associated with a poor prognosis. TGFa and EGF, the ligands for EGFR, are also overexpressed in some of these tumor types, suggesting a self-propagating stimulus that may be responsible for rapid tumor growth. Blocking this stimulus by blocking activation of EGFR with ABX-EGF, a fully human monoclonal antibody against EGFR, may prevent tumor growth and perhaps shrink tumors. Purpose: This is a Phase 2 clinical trial to evaluate the safety and efficacy of ABX-EGF in combination with paclitaxel and carboplatin in the treatment of advanced NSCLC.

ELIGIBILITY:
For complete inclusion and exclusion criteria, please refer to the investigator. Inclusion Criteria: - 18 years of age or older. - Pathological diagnosis of NSCLC. - Bidimensionally measurable disease. - Tumor tissue available for immunohistochemistry studies. - Tumor over-expressing EGFR as ascertained by immunohistochemistry. - Disease stage IIIB with pericardial or pleural effusion, or stage IV. - Life expectancy of at least 12 weeks. - Adequate hematology function - Adequate renal function - Adequate hepatic function - ECOG score of less than 2. - Brain metastases, if present; must be controlled and asymptomatic. Exclusion Criteria: - Calcium > ULN (treatment for hypercalcemia allowed). - Use of any investigational therapy within 30 days of ABX-EGF infusion. - Any cancer therapy for NSCLC other than radiation therapy, surgery, or steroids. - Radiation therapy within 2 weeks before ABX-EGF infusion. - LVEF less than 45% as measured by MUGA. - Symptomatic ventricular arrhythmia or symptomatic conduction abnormality. - Myocardial infarction within 1 year before first dose of study drug. - History of cancer that has required treatment or been active within past 5 years, other than NSCLC, basal cell carcinoma, or cervical carcinoma in situ. - Women (e.g., of childbearing potential, who are post-menopausal for less than six months, not surgically sterilized or not abstinent) who are not willing to use an oral or implanted contraceptive, double barrier birth control, or an IUD during the course of the study and for 6 months following treatment. - Men not willing to use contraception upon enrollment into this study and for 1 month following treatment. - Women who are breast-feeding or have a positive pregnancy test within 72 hours of first study drug administration. - Known to be HIV positive. - Any patient who's best medical interests would not be met by entry in the study in the opinion of the Investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194
Dates: Start 2002-01

PRIMARY OUTCOMES:
Time to Disease Progression

SECONDARY OUTCOMES:
Best Overall Response Rate
Response Rate at Week 5
Survival Time
Progression Free Survival
Rate of Progressive Disease at Week 11
Incidence of AEs
Lab Abnormalities and other Safety Parameters
PK of Panitumumab in Combination with Carboplatin and Paclitaxel
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com